CLINICAL TRIAL: NCT01851551
Title: A Phase I/II Study of Rituximab Plus Vincristine Sulfate Liposomes Injection in the Treatment of Relapsed or Refractory Aggressive Non Hodgkin's Lymphoma
Brief Title: Phase 1/2 Study of VSLI Plus Rituximab in Patients With Relapsed and/or Refractory NHL
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Acrotech Biopharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA00005
Record Dates: First submitted 2013-04-29; First posted 2013-05-10 (Estimated); Last update posted 2020-01-03 (Actual); Status verified 2019-12

CONDITIONS: Non-Hodgkin's Lymphoma; Diffuse Large B-cell Lymphoma; Mantle Cell Lymphoma
Keywords: NHL; non-Hodgkin's lymphoma; diffuse large b-cell lymphoma; mantle cell lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Mantle-Cell | interventions — Rituximab; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VSLI plus rituximab (Experimental): VSLI (vincristine sulfate liposome injection) plus rituximab
  Interventions: Drug: Vincristine Sulfate Liposome Injection plus rituximab

INTERVENTIONS:
Drug: Vincristine Sulfate Liposome Injection plus rituximab
  Other Names: Marqibo; VSLI; rituximab; rituxan

SUMMARY:
This was a Phase 1/2 study performed at two clinical centers in the US and UK. It was a single arm, open label study evaluating VSLI plus rituximab in adults with aggressive relapsed or refractory non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
The primary efficacy endpoint was objective response rate, defined as the proportion of patients with a response of CR + PR.

Duration of response, time to progression, and overall survival were analyzed. Descriptive statistics were used for demographics, disease characteristics, treatment exposures, efficacy, and safety variables.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed diffuse large B-cell non-Hodgkin's lymphoma (NHL), as defined by the Revised European American Lymphoma/WHO classification. This included: diffuse large B-cell, primary mediastinal large B-cell lymphoma with sclerosis,intravascular large B-cell lymphoma, immunoblastic B-cell lymphoma, T-cell rich B-cell lymphoma or anaplastic large B-cell lymphoma. In the US protocol only, patients who had transformation from an indolent lymphoma and those who had mantle cell lymphoma were eligible.

  * Confirmation of CD20 expression on lymphoma cells.
  * Eastern Cooperative Oncology Group (ECOG) ≤2.
  * One or more prior chemotherapy regimens. Patients who had received prior rituximab therapy as part of an induction chemotherapy regimen or who had a previous response to rituximab as a single agent were eligible.
  * Measurable disease in at least 1 site, which had not been previously irradiated.

Measurable disease was defined as at least 1 bidimensionally measurable lesion with clearly defined margins that were ≥1.5 cm in the largest dimension determined by physical examination or computed tomography (CT) scan.

* Total bilirubin and serum creatinine ≤2 times the ULN.
* Absolute neutrophil count (ANC) ≥0.5 × 109/L, and platelets ≥50 × 109/L.
* 18 years of age or older.
* Women of childbearing potential who were willing to use an acceptable method of contraception throughout the course of the study.

Signed and dated informed consent form.

Exclusion Criteria:

* Known transformation from an indolent lymphoma (UK protocol only).
* Eligible for conventional or high-dose chemotherapy with curative intent.
* Radiotherapy, chemotherapy, immunotherapy, or corticosteroids (>10 mg/day of prednisone or equivalent) within the past 4 weeks.
* Any previous malignancies with less than a 5-year complete remission interval, except for curatively resected basal cell carcinoma or curatively resected in situ carcinoma of the uterine cervix.
* History of or active CNS-lymphoma, AIDS-related lymphoma, or any uncontrolled severe medical illness or infection.
* History of neurologic disorders unrelated to chemotherapy (including familial neurologic diseases and acquired demyelinating disorders).
* Grade 3 or 4 sensory or motor neuropathy at screening related to prior chemotherapy.
* Major surgery (excluding that for diagnosis) within 4 weeks of enrollment.
* Pregnant or lactating women (women of childbearing potential underwent a pregnancy test).
* Allergy to vincristine, or other vinca alkaloids.
* Progressive disease while receiving or within 1 month of having received previous rituximab therapy (US protocol only).
* Hypersensitivity to any component of rituximab or to murine proteins (UK protocol only).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2001-09; Primary Completion 2004-04 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Objective response rate | Assessed prior to each cycle for up to 12 cycles (24 weeks). For patients achieving a complete or partial response, follow-up assessments were to be made 2, 8, 16, and 24 weeks after treatment was discontinued (up to ~48 wks).
  The primary efficacy endpoint was the objective response rate (ORR) defined as the proportion of patients whose best responses were complete response (CR) and partial response (PR) (ORR = CR + PR).

SECONDARY OUTCOMES:
Assessment of the number of events and number and percentage of patients with treatment-emergent AEs | AEs were assessed up to 30 days post last dose. Dosing may last up to 24 weeks.
  The number of events and number and percentage of patients with treatment-emergent AEs that occurred from the time of first study treatment up to 30 days following the last study treatment were summarized by MedDRA system organ class and preferred term, NCI CTC grade, and relationship to study drug.
  Safety variables included adverse events, neurologic assessments, chemistry and hematology laboratory tests, physical examinations, and vital signs.
  Neurologic symptom scores were summarized for baseline and worst score on study. The number and percentage of patients with neurologic symptom abnormalities were tabulated and presented by severity and cycle for each symptom.
  Neurologic sign scores were summarized for baseline and worst score on study. The number and percentage of patients with neurologic sign abnormalities were tabulated and presented by severity and cycle for each sign.
  Shifts from baseline to worst value were tabulated by cycle based on NCI CTC grades
Time to Progression | First dose to disease progression. Follow up was reported approximately every 3 months post-dose up to the date of patient death. Patients were followed up to 2 yrs.
  Time To Progression (TTP), defined as the interval between the initial day of dosing and disease progression or death due to NHL
Overall survival | The interval between first dose and death due to any cause. Reported every 3 months post dose up to patient death. Follow up was approximately 2 years
  Overall Survival (OS) was defined as the interval between the initial day of dosing and death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Kaplan, MD, Principal Investigator — University of California, San Francisco; Gareth Morgan, Prof., Principal Investigator — Leeds General Infirmary
Locations (2):
- University of California, San Francisco, California, United States
- Leeds General Infirmary, Leeds, West Yorkshire, United Kingdom